CLINICAL TRIAL: NCT06607081
Title: The Preoperative Risk Evaluation and Perioperative ERAS Intervention in the Chinese Elderly Patients Underwent Spinal Fusion Surgery
Brief Title: Preoperative Risk Evaluation and Per ERAS Intervention in the Chinese Elderly Patients Underwent Spinal Fusion Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Shenzhen Hospital of Southern Medical University (Other); Second Xiangya Hospital of Central South University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20242310wuzixiang
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Degenerative Spinal Disease; Elderly Patients; Spinal Fusion Acquired
Keywords: Elderly patients; ERAS; Spinal disease; Surgical intervention; Risk factors
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perioperative Pre ERAS group (Experimental)
  Interventions: Combination Product: Multidisciplinary Preoperative Risk Evaluation and the Corresponded Pre ERAS intervention
- Control group (No Intervention)

INTERVENTIONS:
Combination Product: Multidisciplinary Preoperative Risk Evaluation and the Corresponded Pre ERAS intervention — The operative risk factors are multidisciplinary evaluated and the corresponded multimodal measures are used to optimize the whole condition of the elderly patient undergo spinal fusion surgery for his/her safty, early and fully recovery.
  Arms: Perioperative Pre ERAS group

SUMMARY:
This study aims to evaluate the value of preoperative risk factor evaulation combined with perioperative ERAS measures in improving the clinical prognosis of elderly patients undergo the spinal fusion.

DETAILED DESCRIPTION:
Population ageing is rapid progressing globally. In the United States, the number of people over the age of 80 is expected to grow from 1.9% in 2020 to 4.3% in 2050. According to the Statistical Communique on the Development of Civil Affairs in 2023 issued by the Ministry of Civil Affairs in 2024, the elderly population aged 65 and above in China is 216.76 million, accounting for 15.4% of the total population. Spinal degenerative diseases are the most common diseases among the elderly population. The prevalence of spinal degenerative diseases over 65 years old is about 56%, and there are about 121 million patients in China. Spinal degenerative diseases, including cervical spondylosis, cervical spinal stenosis, lumbar disc herniation, lumbar spinal stenosis, degenerative scoliosis, et al., which can lead to significant nerve compression, pain, neurological dysfunction, and mobility and endurance reduction, leading to reduced quality of life. Elderly patients preferentially choose non-surgical treatment such as drug intervention, but most conservative treatment methods have limited efficacy and cannot completely relieve nerve compression. Spinal fusion surgery is the most fundamental solution to the treatment of spinal degenerative diseases. Because of the elderly patients with multiple diseases, multi-drug use, multi-organ dysfunction, therefore, the perioperative safety management of such patients is a difficult problem faced by clinicians.

Preoperative high-risk factor evaluation and pre-enhanced recovery after surgery (Pre ERAS) are effective preoperative optimization strategies to benefit elderly patients. Patients are comprehensively evaluated before surgery by multidisciplinary consultation group to assess the high risk factors of spinal fusion surgery. On this basis, multidisciplinary intervention, exercise, nutritional support and psychological intervention were carried out to increase patients' preoperative physiological reserve, reduce the incidence of postoperative adverse events, and ultimately improve patients' perioperative functional status and prognosis. However, there is still a significant lack of unified understanding and willingness to implement preoperative screening and surgical management for elderly patients.

On the basis of "Chinese Expert Consensus on Multidisciplinary Evaluation of Perioperative Period in Elderly Spinal Surgery Patients", this study intends to further specify the concept of Pre ERAS for diagnosis and treatment measures, and form an operable Pre ERAS protocol. Through multi-center, prospective clinical study, to comprehensively evaluate the comprehensive impact of preoperative high-risk factor assessment combined with Pre ERAS measures on the clinical prognosis of elderly patients undergoing spinal fusion surgery, which lays an evidence-based medical foundation for the extensive application of this concept and measures in clinical practice.

The overall aim of this work is to evaluate the effects of preoperative risk factors and Pre ERAS on clinical outcomes in elderly (≥75 years) spinal fusion patients.

This study is a multi-center, prospective, randomized controlled clinical trial including a total of 2500 patients in the experimental group and the control group, respectively. The research centers include: Shenzhen Hospital of Southern Medical University, the Second Xiangya Hospital of Central South University, and Shanghai General Hospital. Patients were recruited according to inclusion criteria and exclusion criteria. The experimental group received Pre ERAS during perioperative period, while the control group received conventional ERAS during perioperative period. According to the clinical study protocol, patients were subjected to perioperative intervention, clinical follow-up, results recorded, adverse events were discovered and recorded in time and reported according to regulations, and cases meeting the exclusion criteria were excluded. This study will start in October 2024. The recruitment period will be 12 months, with a follow-up of 12 months. The results of the study will be expected in October 2027.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥75 years old;
* 2.Have degenerative spinal diseases, including cervical, thoracic and lumbar spine diseases;
* 3.With severe neurological symptoms fail to conservative treatment and have to undergo the spinal fusion surgery;
* 4.No serious cognitive impairment (MoCA score ≥8);
* 5.No surgical contraindications;
* 6.Anesthesia assessment patients can safely undergo surgery;
* 7.Patients who voluntarily participate in and sign informed consent, can independently complete effective questionnaires, and are willing to follow up according to clinical requirements.

Exclusion Criteria:

* 1.Patients who could not cooperate with doctors to complete preoperative evaluation and postoperative follow-up;
* 2.Patients requiring spinal intervention due to spinal infection, fracture or metastatic disease;
* 3.Patients with cerebrovascular accidents in the last 30 days;
* 4.Patients with hepatic encephalopathy or acute active hepatitis;
* 5.Patients with severe renal insufficiency with creatinine>2.5mg/dL or undergoing hemodialysis;
* 6.Patients with severe lung and cardiovascular diseases, coagulation disorders, and anesthesia contraindications;
* 7.Patients with poorly controlled diabetes (HBAlc>8.0%);
* 8.Patients who are participating in clinical trials of other drugs or medical devices;
* 9.Patients requiring emergency surgery;
* 10.Patients who are considered by the investigator to be unable to participate in this clinical trial due to other circumstances.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Complication Index | 24 weeks postoperation
  The Comprehensive Complication Index (CCI) is based on the complication grading by the Clavien-Dindo Classification and captures every complication that occurred after an intervention. The overall morbidity is reflected on a scale from 0 (no complication) to 100 (death) and reflects the gravity of this overall complication burden on the patients. CCI can be calculated using online CCI calculator (https://cci-calculator.com/cciCalculator), which is a tool to support the assessment of patients' overall morbidity after an intervention.

SECONDARY OUTCOMES:
Neck disability index (NDI) score/Oswestry disability index (ODI) score | 24 weeks postoperation
  The Neck disability index (NDI) score reflects the neck-related functional status of patients with cervical spine pathology and response to the surigcal treatment. The NDI score is assessed using NDI questionnaire and the total NDI score ranges from 0 to 50 points, with the highest socre (50 pionts) means complete disability and the lowest socre (0 points) means no disability.
  The Oswestry disability index (ODI) score reflects back-related functional status of patients with lumbar spine pathology and response to the surgical treatment. The ODI score is assessed using ODI questionnaire. The total ODI score is reported from 0 to 100, with the higher score reflects higher disability and lower functional status, while the lower score reflects lower disability and higher functional status.
North American Spine Satisfaction (NASS) Score | 24 weeks postoperation
  The patient satisfaction after spinal fusion intervention is assessed using North American Spine Satisfaction (NASS) questionnaire. NASS score ranges from 1 to 4, the lowest score means the highest level of satisfication while the highest score means the lowest level of satisfication.
  Score 1 is defined as "Surgery met my expectations." Score 2 is defined as "I did not improve as much as I had hoped but I would undergo the same operation for the same results." Score 3 is defined as "Surgery helped but I would not undergo the same operation for the same results," Score 4 is defined as "I am the same or worse as compared to before surgery."
Japanese Orthopaedic Association (JOA) score | 24 weeks postoperation
  The severity of cervical compression myelopathy before and after surgery of the patients is evaluated using the Japanese Orthopaedic Association (JOA) scale, with the total JOA score ranges from 0 to 17. If the JOA score is larger than 13, the severity defines as mild. If the JOA score is 9~13, the severity defines as moderate. If the JOA score is less than 9, the severity defines as severe.
Bone minral density (BMD) evaluation | 24 weeks postoperation
  The bone minral density (BMD) will be tested using Dual Energy X-ray Absorptiometry (DEXA) to assess the bone quality of the patients included in this study before and after spinal fusion intervention.
Spinal fusion rates | 24 weeks postoperation
  The spinal fusion is evatluted by compute tomography (CT) scanning to reflects the effectiveness of Pre ERAS on bone healing after surgical intervention.
  The spinal fusion criteria is defined as the continuous callus is detected on CT radiograph at the surgical intervented spinal segments.
  The spinal fusion rates is calculated as the number of the fused setgments after surgical intervention divided by the number of the total surgical intervented segments.
Length of hospital stay | 2 weeks postoperation
  The length of hospital stay is the total time of the patient spended in hospital for medical treatment. This time starts from patient admission and ended when patient discharge.
  The discharge criteria:
  1. The patient satified with the outcomes of spinal fusion intervention;
  2. The spinal fusion intervention achieved peroperative symptoms relive and function recovery;
  3. No further medical intervention is needed;
  4. No surgerical complications;
Discharge rate | 2 weeks postoperation
Readmission rate | 4 weeks postoperation
90-day unplanned readmission rates | 90 days postoperation
  Any admission which was within 90 days of the previous discharge (index admission) was counted as 90-day unplanned readmission.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chotai S, Devin CJ, Archer KR, Bydon M, McGirt MJ, Nian H, Harrell FE Jr, Dittus RS, Asher AL; QOD Vanguard Sites. Effect of patients' functional status on satisfaction with outcomes 12 months after elective spine surgery for lumbar degenerative disease. Spine J. 2017 Dec;17(12):1783-1793. doi: 10.1016/j.spinee.2017.05.027. Epub 2017 Sep 29. PMID 28970074
- [Background] Kim TI, Brahmandam A, Skrip L, Sarac T, Dardik A, Ochoa Chaar CI. Surgery for the Very Old: Are Nonagenarians Different? Am Surg. 2020 Jan 1;86(1):56-64. PMID 32077417
- [Background] Kim DU, Park HK, Lee GH, Chang JC, Park HR, Park SQ, Cho SJ. Central Sarcopenia, Frailty and Comorbidity as Predictor of Surgical Outcome in Elderly Patients with Degenerative Spine Disease. J Korean Neurosurg Soc. 2021 Nov;64(6):995-1003. doi: 10.3340/jkns.2021.0074. Epub 2021 Oct 7. PMID 34614555
- [Background] Carlstrom LP, Helal A, Perry A, Lakomkin N, Graffeo CS, Clarke MJ. Too frail is to fail: Frailty portends poor outcomes in the elderly with type II odontoid fractures independent of management strategy. J Clin Neurosci. 2021 Nov;93:48-53. doi: 10.1016/j.jocn.2021.08.027. Epub 2021 Sep 11. PMID 34656260
- [Background] Debono B, Corniola MV, Pietton R, Sabatier P, Hamel O, Tessitore E. Benefits of Enhanced Recovery After Surgery for fusion in degenerative spine surgery: impact on outcome, length of stay, and patient satisfaction. Neurosurg Focus. 2019 Apr 1;46(4):E6. doi: 10.3171/2019.1.FOCUS18669. PMID 30933923
- [Background] van Rooijen S, Carli F, Dalton S, Thomas G, Bojesen R, Le Guen M, Barizien N, Awasthi R, Minnella E, Beijer S, Martinez-Palli G, van Lieshout R, Gogenur I, Feo C, Johansen C, Scheede-Bergdahl C, Roumen R, Schep G, Slooter G. Multimodal prehabilitation in colorectal cancer patients to improve functional capacity and reduce postoperative complications: the first international randomized controlled trial for multimodal prehabilitation. BMC Cancer. 2019 Jan 22;19(1):98. doi: 10.1186/s12885-018-5232-6. PMID 30670009
- [Background] Soffin EM, Beckman JD, Tseng A, Zhong H, Huang RC, Urban M, Guheen CR, Kim HJ, Cammisa FP, Nejim JA, Schwab FJ, Armendi IF, Memtsoudis SG. Enhanced Recovery after Lumbar Spine Fusion: A Randomized Controlled Trial to Assess the Quality of Patient Recovery. Anesthesiology. 2020 Aug;133(2):350-363. doi: 10.1097/ALN.0000000000003346. PMID 32433277